CLINICAL TRIAL: NCT06541171
Title: A New Fast DWI-based Magnetic Resonance Protocol for Surveillance in Patients With a High Risk of Ovarian Cancer Recurrence During PARP-inhibitors Maintenance to Enhance Secondary Cytoreduction Results
Brief Title: A New Fast DWI-based MR Protocol for Surveillance in Patients With a High Risk of Ovarian Cancer Recurrence During PARP-inhibitors Maintenance to Enhance Secondary Cytoreduction Results
Acronym: FOFU
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6887
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Ovarian Cancer; Recurrent Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Magnetic resonance imaging as fpr clinical practice — An abbreviated MR protocol of the abdomen will be used inh association with CT scan; it does not need contrast injection and does not add any risk for patients.

SUMMARY:
In ovarian cancer (OC), complete surgical debulking and platinum-based chemotherapy are the standard treatment, now followed by maintenance therapy with PARP inhibitors or Bevacizumab. However, in advanced-stage ovarian cancer, recurrence is common, with a progression-free survival of about 16 months. Secondary cytoreductive surgery (SCS) at the time of recurrence prolongs the overall survival and gives the possibility to extend the use of PARP-i. SCS is possible only when recurrence has limited extension. However, in OC, there is no well-established and widely accepted scheme for surveillance during maintenance therapy; ESMO guidelines suggest physical examination for the follow-up and allow ultrasound, CT, PET-CT and MRI to confirm the recurrence and plan surgical treatment if appropriate.

DETAILED DESCRIPTION:
Patients with OC in surveillance after first-line treatment usually have a scheme of clinical visits and serum marker evaluation every three months, associated with alternated transvaginal ultrasound and chest, abdomen and pelvis CT with contrast every three months and MRI with a confirmatory role in some cases.

We will use an abbreviated MR protocol of the abdomen (the most common location of relapse and the only one that can be treated by surgery) in association with CT. The abbreviated protocol is based on axial b50, b600 and b900 DWI with three-dimensional coronal maximum intensity projection (MIP) reconstruction of b900 values, ADC maps and axial single-shot T2-weighted sequences, which will take less than 20 minutes. This MRI protocol does not need contrast injection and does not add any risk for patients.

Any positive findings will be discussed at the Multidisciplinary Tumour Board and secondary cytoreductive surgery will be evaluated. Surgery outcome and subsequent clinical information (secondary PFS and OS) derived by normal clinical practise will be registered in a dedicated database.

ELIGIBILITY:
Inclusion Criteria:

* Patients with BRCA wild-type, HRP, high-grade serous ovarian cancer
* No residual tumour at first debulking surgery
* More than 6 months since the last platinum-based therapy

Exclusion Criteria:

* Patients who will not consent to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of HGSOC with BRCA wild-type, without residual tumour after first debulking surgery, who are planned for CT/MRI exams as for Follow Up Clinical Practice, after more than 6 months since the last platinum-based therapy
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Cytoreductive surgery rate | 36 months
  Optimal cytoreductive surgery rate

SECONDARY OUTCOMES:
Concordance rate between MRI results and CA125 variations | 36 months
  Percentage of Concordance between MRI results and CA125 variations
Concordance between MRI results and CT findings | 36 months
  Percentage of Concordance between MRI results and CT findings
Rate of Survival | 36 months
  Progression-Free Survival and Overall Survival Rate

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Avesani, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitaro "A. Gemelli" IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No